CLINICAL TRIAL: NCT05251558
Title: The Efficacy of Telerehabilitation Based Self Proprioceptive Neuromuscular Facilitation Exercises on Clinical and Psychosocial Parameters in Bell's Palsy Patients
Brief Title: Efficacy of Telerehabilitation Based Exercises in Patients With Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BELLS1
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bell Palsy
Keywords: Bells Pasly; Telerehabilitation; Peripheral Facial Paralysis; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Bell Palsy; Facial Paralysis | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) (Experimental): Self PNF exercises determined for facial muscles (M. Frontalis, M. Orbicularis Oculi, M. Orbicularis Oris, M. Risorius etc.) will be applied.
  Interventions: Other: Telerehabilitation
- Conventional Education Program (CEP) (Active Comparator): Education will be given to cases with Bell's Palsy. Some exercises will be suggested in front of the mirror. Patients will be advised to gently massage upwards with their fingertips after applying a warm towel with a towel on the facial muscles.
  Interventions: Other: Conventional Education Program

INTERVENTIONS:
Other: Telerehabilitation — The telerehabilitation platform is used to deliver the home exercise program.
  Arms: Telerehabilitation (TR)
Other: Conventional Education Program — The patient is given education about the points to be considered for the disease and the exercises to be applied.
  Arms: Conventional Education Program (CEP)

SUMMARY:
The study will be carried out with volunteer patients who are diagnosed with Bell's Palsy and comply with the study criteria.The aim of the study is to compare the home PNF exercise program with video-based telerehabilitation and the conventional training program in terms of outcome measures in patients with Bell's Palsy lesions.

DETAILED DESCRIPTION:
With the telerehabilitation program, it is aimed that patients can easily adapt to home exercise programs and be followed up remotely. In this way, the most effective treatment of the disease will provide the patient with both motor function gain and psychosocial gain. This study was planned to examine the effectiveness of telerehabilitation in patients with Bell's Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 65 years
* Being diagnosed with Bell's Palsy by a specialist physician
* Having a lower motor neuron lesion
* Non-traumatic cases
* Not having any other neurological deficits
* Having signed the consent form

Exclusion Criteria:

* Situations that will prevent assessments or communication with the individual
* Bilateral involvement
* Having an operation for facial palsy
* Having an upper motor neuron lesion
* Neurological problems that would preclude evaluation and/or treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
FDI | Change from Baseline FDI at 4 weeks
  The Facial Disability Index is a questionnaire that provides information about the impact of facial paralysis and the physical and social well-being impairment it causes. FDI is scored from 0 to 100. Higher scores indicate better function.
FaCE | Change from Baseline FaCE at 4 weeks
  It consists of 15 items with responses on a 5-point Likert scale in 6 sub-categories: facial movements, social function, facial comfort, tear control, eye comfort, and mouth function. FaCE is scored from 0 to 100. Higher scores indicate better function.
SF-12 | Change from Baseline SF-12 at 4 weeks
  SF 12 is a self-evaluation scale. It consists of seven items. SF-12 is scored from 0 to 100. Higher scores indicate better quality of life.
HADS | Change from Baseline HADS at 4 weeks
  The scale includes anxiety and depression subscales. The purpose of the scale is not to diagnose, but to determine the risk group by scanning anxiety and depression in a short time in patients with physical illness. HADS is scored from 0 to 21. Higher scores indicate higher depression and anxiety.
H-B | Change from Baseline H-B at 4 weeks
  The scale evaluates the four facial regions separately and also assesses the presence of synkinesis. H-B is scored from 4 to 24. Higher scores indicate worse clinical status.

SECONDARY OUTCOMES:
TSUQ | Change from Baseline TSUQ at 4 weeks
  With this survey, the satisfaction levels and usability of individuals using the telemedicine service are evaluated. TSUQ is scored from 21 to 105. Higher scores indicate higher satisfaction and usability.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University; Mehmet Özkeskin, PhD, Principal Investigator — Ege University; İsmet Tümtürk, MSc, Principal Investigator — Süleyman Demirel University; Yalçın Gölcük, MD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sıtkı Kocman University Hospital Emergency Service, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No